CLINICAL TRIAL: NCT00531947
Title: A Phase IV, Double-Blind, Placebo-Controlled, Randomized, Flexible Dose Study of the Safety and Efficacy of EMSAM in Adolescents With Major Depression
Brief Title: Phase IV:Safety and Efficacy of EMSAM in Adolescents With Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Somerset Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S9303-P0605
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Mental Health; Adolescents; Major Depressive Disorder; Depression; Adolescent Depression; Pediatric Depression
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMSAM (Experimental): Approved Medication for Major Depressive Disorder: EMSAM (Selegiline Transdermal System) 6mg, 9mg, or 12mg
  Interventions: Drug: Selegiline Transdermal System
- Placebo (Placebo Comparator): Placebo Selegiline Transdermal System 6, 9 or 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selegiline Transdermal System — EMSAM 6mg, 9mg, or 12mg Flexible Dose- 1 patch/24 hours- 12 Week Study
  Other Names: EMSAM
  Arms: EMSAM
Drug: Placebo — Matching Placebo for EMSAM 6mg, 9mg, or 12mg Flexible Dose- 1 patch/24 hours- 12 Week Study
  Other Names: Matching Placebo Transdermal System
  Arms: Placebo

SUMMARY:
The primary purpose of your participation in this study is to help answer the following research question: Whether 12-week administration of EMSAM (selegiline transdermal system) is safe and effective for the treatment of adolescents (aged 12 through 17 years) with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
• Assess the safety and efficacy of EMSAM (selegiline transdermal system) versus placebo in adolescents (aged 12 through 17 years) who meet criteria for Major Depressive Disorder (MDD) without psychotic features, single or recurrent

ELIGIBILITY:
Inclusion Criteria:

* Male / Female outpatients 12 to 17 years of age diagnosed with Major Depressive Disorder (MDD). (Must have a Children's Depression Rating Scale-Revised [CDRS-R] with a total score of at least 45 at screening.)
* Female patients must test negative on a pregnancy at visit 1.
* Weight and height must be greater than the 10th percentile according to age and height,
* Assent and consent must be given.

Exclusion Criteria:

* Have a serious or unstable medical illness, psychological condition, clinically significant laboratory or ECG result, hypersensitivity to selegiline, or any other condition that in the opinion of the investigator would compromise participation in the study or be likely to lead to hospitalization during the course of the study.
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, pervasive development disorder or borderline personality disorder, as determined by the investigator.
* Have a risk of suicide
* Female patients who are either pregnant, nursing or have recently given birth.
* Use of any protocol prohibited medications or substances.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 308 (Actual)
Dates: Start 2007-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hochadel, Pharm.D., Study Director — Cognitive Research Corporation; Melissa L Goodhead, Study Chair — Somerset Pharmaceuticals
Locations (20):
- United States (20):
  - Dr. Nelson Handal, Dothan, Alabama
  - Dr. Mohammed Bari, National City, California
  - Dr. Michael McManus, San Diego, California
  - Dr. Elias Sarkis, Gainesville, Florida
  - Dr. Scott Segal, North Miami, Florida
  - Dr. Mary Stedman, Tampa, Florida
  - Dr. Irving Kolin, Winter Park, Florida
  - Dr. Rory Murphy, Overland Park, Kansas
  - Dr. Andrew Sediloo, Owensboro, Kentucky
  - Dr. Bruce Waslick, Springfield, Massachusetts
  - Dr. Christopher Kratochvil, Omaha, Nebraska
  - Dr. Ann Childress, Las Vegas, Nevada
  - Dr. Melissa DelBello, Cincinnati, Ohio
  - Dr. Leland Dennis, Oklahoma City, Oklahoma
  - Dr. David Brown, Austin, Texas
  - Dr. Alain Katic, Bellaire, Texas
  - Dr. Graham Emslie, Dallas, Texas
  - Dr. Mary Shemo, Charlottesville, Virginia
  - Dr. John Gilliam, Richmond, Virginia
  - Dr. Arifulla Khan, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female adolescent subjects between 12 to 17 years of age diagnosed with moderate to severe major depressive disorder were screened over an approximate two year period at 26 investigative sites in the U.S.
Groups:
- Placebo: Placebo Selegiline Transdermal System 6, 9 or 12
  Placebo : Matching Placebo for EMSAM 6mg, 9mg, or 12mg Flexible Dose- 1 patch/24 hours- 12 Week Study
- EMSAM: Approved Medication for Major Depressive Disorder: EMSAM (Selegiline Transdermal System) 6mg, 9mg, or 12mg
  Selegiline Transdermal System : EMSAM 6mg, 9mg, or 12mg Flexible Dose- 1 patch/24 hours- 12 Week Study
Period: Overall Study
Arm/Group | Placebo | EMSAM
Started | 156 (all randomized subjects who received at least one dose of placebo study medication) | 152 (all randomized subjects who received at least one dose of EMSAM study medication)
Completed | 114 | 101
Not Completed | 42 | 51
Not completed — Adverse Event | 5 | 10
Not completed — Lost to Follow-up | 12 | 9
Not completed — Withdrawal by Subject | 14 | 19
Not completed — Protocol Violation | 2 | 1
Not completed — Non-Compliance | 4 | 7
Not completed — Other (e.g., Lack of Efficacy) | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EMSAM | Total
Number analyzed (Participants) | 156 | 152 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 156 | 152 | 308
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6) | 14.8 (1.62) | 14.8 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 93 | 197
  Male | 52 | 59 | 111
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 77 | 69 | 146
  Black | 34 | 46 | 80
  Hispanic | 37 | 32 | 69
  Asian | 2 | 1 | 3
  Native American | 1 | 1 | 2
  Other | 5 | 3 | 8

OUTCOME MEASURES:

1. Secondary Outcome: CGI-S - Week 12 (mITT w/LOCF Population)
Description: A summary of the Clinical Global Impression of Severity (CGI-S) at baseline and Week 12 (EOS), by treatment assigned, is shown for the mITT population with LOCF. The CGI-s is the clinician's assessment of severity of illness (depression). Scores range from 1(minimum) to 7(maximum). A lower score indicates lower illness severity, a higher score indicates higher levels of illness severity.
Time Frame: Baseline and 12 Weeks
Population: Received at least one dose of placebo or EMSAM study drug, and had at least one post-treatment efficacy assessment with the primary outcome variable (CDRS-R).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 150
units on a scale
  Baseline CGI-S Scale | 4.494 (0.659) | 4.527 (0.662)
  Week 12 CGI-S Scale | 3.000 (1.333) | 3.007 (1.250)

2. Secondary Outcome: CGI-C - Week 12 (mITT w/LOCF Population)
Description: A summary of the Clinicians Global Impression of Change (CGI-C) Score at Week 12 (EOS), by treatment assigned, is shown for the mITT population with LOCF. The CGI-c assesses the overall change in the severity of illness (depression). The clinician rates the subject's change based on a bipolar scale from 1(minimum; "Very much improved") to 7(maximum; "Very much worse"). A lower score indicates lower levels of depression as compared to baseline, a higher score indicates higher levels of depression as compared to baseline. A score of 4 ("Unchanged") indicates no change in illness compared to baseline. The scale is not calculated as a statistical change score; the clinician rates their impression of change overall.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 150
units on a scale | 2.387 (1.208) | 2.386 (1.138)

3. Secondary Outcome: CGI-C Percent Responders (mITT w/LOCF Population)
Description: A summary of the CGI-C percent responders at Week 12 (EOS), by treatment assigned, is shown for the mITT population with LOCF. CGI-C responders were defined as a score of 1 or 2 at the end of the study. A non-responder was defined as a score of ≥3 at end of study. Maximum score is 100%.
Time Frame: 12 Weeks
Measure: Number; unit: Percent Responder
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 150
Percent Responder
  Percent Non-Responder | 40.7 | 41.4
  Percent Responder | 59.3 | 58.6

4. Secondary Outcome: CDRS-R Total Score (Parent/Other) Week 12 (mITT w/LOCF Population)
Description: A summary of a secondary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score (Scored by Parent/Other), at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population, with the last observation carried forward (LOCF) in time.
  CDRS-R (Parent/Other) total raw scores range from 14 (minimum) 94 (maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. One subscale is summed to calculate a total score: Evaluated Symptom Area. Ratings of Observed Nonverbal Behavior subscale is not included in Parent/Other total calculation.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 149
units on a scale
  Baseline- Observed | 49.4 (11.27) | 48.8 (10.1)
  Week 12- Observed | 30.7 (13.55) | 30.5 (13.36)
  Week 12 - Change From Baseline | -18.7 (14.09) | -18.3 (14.27)

5. Secondary Outcome: CDRS-R Total Score (Best Description) Week 12 (mITT w/LOCF Population)
Description: A summary of a secondary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score (Best Description), at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population, with the last observation carried forward (LOCF) in time.
  Best Description ratings are used when ratings based on interviews with different sources (e.g., child, parent, other ratings) differ for a particular symptom. The evaluator must determine which of these ratings most accurately represents the current affective functioning of the child, and circle that rating in the Best Description of Child Column.
  CDRS-R (Best Description)total raw scores range from 17(minimum) 113(maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. Two subscales are summed to calculate a total score: Evaluated Symptom Area and Ratings of Observed Nonverbal Behavior.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 150
units on a scale
  Baseline - Observed | 60.7 (12.26) | 59.5 (11.05)
  Week 12 - Observed | 38 (16.62) | 37 (15.73)
  Week 12 - Change From Baseline | -22.7 (16.54) | -22.5 (16.97)

6. Secondary Outcome: CDRS-R Total Score (Child) Week 12 (mITT w/OC Population)
Description: A summary of the secondary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score (Scored by Child), at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population with observed cases (w/OC).
  CDRS-R (Child) total raw scores range from 17(minimum) 113(maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. Two subscales are summed to calculate a total score: Evaluated Symptom Area and Ratings of Observed Nonverbal Behavior.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 151 | 146
units on a scale
  Baseline - Observed | 58.1 (12.64) | 56.6 (12.39)
  Week 12 - Observed | 30.8 (12.41) | 31.1 (12.38)
  Week 12 - Change From Baseline | -25.5 (15.07) | -25.3 (15.16)

7. Secondary Outcome: CDRS-R Total Score (Parent/Other) Week 12 (mITT w/OC Population)
Description: A summary of a secondary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score (Scored by Parent/Other), at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population with observed cases (w/OC).
  CDRS-R (Parent/Other) total raw scores range from 14 (minimum) 94 (maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. One subscale is summed to calculate a total score: Evaluated Symptom Area. Ratings of Observed Nonverbal Behavior subscale is not included in Parent/Other total calculation.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 151 | 146
units on a scale
  Baseline - Observed | 49.6 (11.43) | 48.9 (10.21)
  Week 12 - Observed | 25.5 (10.70) | 25.8 (9.59)
  Week 12 - Change From Baseline | -22.6 (12.97) | -22.2 (12.66)

8. Secondary Outcome: CDRS-R Total Score (Best Description) Week 12 (mITT w/OC Population)
Description: A summary of a secondary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score (Best Description), at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population, with observed cases (w/OC).
  Best Description ratings are used when ratings based on interviews with different sources (e.g., child, parent, other ratings) differ for a particular symptom area. The evaluator must determine which of these ratings most accurately represents the current affective functioning of the child, and circle that rating in the Best Description of Child Column.
  CDRS-R (Best Description) total raw scores range from 17(minimum) 113(maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. Two subscales are summed to calculate a total score: Evaluated Symptom Area and Ratings of Observed Nonverbal Behavior.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 151 | 146
units on a scale
  Baseline - Observed | 60.7 (12.34) | 59.4 (11.10)
  Week 12 - Observed | 32.1 (13.18) | 32.4 (12.75)
  Week 12 - Change From Baseline | -27 (14.93) | -26.6 (15.18)

9. Primary Outcome: CDRS-R Total Score (Child) (mITT w/LOCF Population) Week 12
Description: A summary of the primary efficacy outcome measure, Children's Depression Rating Scale (CDRS-R) Total Score, as reported by the Child, at Week 12 (EOS), by treatment assigned, is shown for the modified intent-to-treat (mITT) population, with the last observation carried forward (LOCF) in time.
  CDRS-R total raw scores range from 17(minimum) 113(maximum). A lower score indicates a lower likelihood of a depressive disorder, a higher score indicates a higher likelihood of a depressive disorder. Two subscales are summed to calculate a total score: Evaluated Symptom Area and Ratings of Observed Nonverbal Behavior.
Time Frame: baseline and 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 154 | 150
units on a scale
  Baseline - Observed | 57.9 (12.57) | 56.7 (12.34)
  Week 12 - Observed | 36.4 (15.91) | 35.4 (15.30)
  Week 12 - Change From Baseline | -21.5 (16.47) | -21.4 (16.61)

10. Secondary Outcome: Physical Examination (Screening vs. EOS)
Description: Number of physical examination findings that were normal at screening, but abnormal at end of study are presented. Four subjects receiving placebo and four subjects receiving EMSAM had abnormal findings on physical examination at the end of study that were normal at screening.
Time Frame: 12 Weeks
Measure: Number; unit: Number of Abnormal Exams
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
Number of Abnormal Exams | 4 | 4

11. Secondary Outcome: Urinalysis (Change From Baseline)
Description: A summary of a secondary safety outcome measure, Urinalysis (Change from Baseline), by treatment assigned, is shown for the safety population. Mean changes from baseline are provided for PH and specific gravity.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
units on a scale
  PH | -0.02 (0.906) | -0.11 (1.052)
  Specific Gravity | 0.00 (0.008) | 0.00 (0.008)

12. Secondary Outcome: Vital Signs-Heart Rate (Change From Baseline)
Description: Summary mean change in heart rate measured in beats per minute (beats/min or BPM) (supine, standing, and orthostatic change)results for all subjects are presented.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 139 | 131
BPM
  Supine Heart Rate | .20 (11.90) | -.10 (9.91)
  Standing Heart Rate | -0.6 (14.26) | 2.6 (15.12)
  Orthostatic Change in Heart Rate | -.80 (11.70) | 2.80 (13.8)

13. Secondary Outcome: Vital Signs-Blood Pressure (Change From Baseline)
Description: Summary mean change in blood pressure (systolic/diastolic) measured in millimeters of mercury (mmHg) (supine, standing, and orthostatic change)results for all subjects are presented.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 139 | 131
mmHg
  Supine Systolic Blood Pressure | 0.9 (8.94) | -0.3 (11.8)
  Supine Diastolic Blood Pressure | 1.1 (8.21) | 1.4 (8.52)
  Standing Systolic Blood Pressure | -1.2 (10.29) | -2.5 (11.63)
  Standing Diastolic Blood Pressure | 0.8 (8.5) | -0.1 (9.11)
  Orthostatic Change in Systolic Blood Pressure | -2.1 (9.32) | -2.3 (11.30)
  Orthostatic Change in Diastolic Blood Pressure | -0.4 (7.84) | -1.5 (7.85)

14. Secondary Outcome: 12 Lead ECG (Change From Baseline)
Description: A summary of a secondary safety outcome measure, 12 Lead electrocardiogram (ECG) (Change from Baseline) measured in milliseconds (msec), by treatment assigned, is shown for the safety population. Mean change from Baseline in PR interval, QRS duration, QT interval, and QTc (Bazett and Fridericia corrections) interval are presented.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
msec
  PR Interval | 0.70 (10.47) | -0.90 (11.04)
  QRS Duration | -0.0 (5.84) | 1.1 (8.21)
  QT Interval | 1.30 (24.86) | 3.80 (21.51)
  QTc (Bazett Correction) Interval | -4.10 (19.20) | -2.90 (20.23)
  QTc (Fridericia Correction) Interval | -2.30 (16.06) | -0.60 (15.27)

15. Secondary Outcome: 12 Lead ECG (Change From Baseline)Ventricular Heart Rate
Description: A summary of a secondary safety outcome measure, 12 Lead electrocardiogram (ECG) (Change from Baseline)Ventricular Heart Rate measured in beats per minute(beats/min or BPM), by treatment assigned, is shown for the safety population. Mean change from baseline is presented.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
BPM | -1.70 (10.40) | -2.40 (10.43)

16. Secondary Outcome: Hematology - White Blood Cell (WBC) (Change From Baseline)
Description: A summary of a secondary safety outcome measure, Hematology (Change from Baseline), by treatment assigned, is shown for the safety population. Mean change from Baseline in ABS BASOPHILS (X10^9/L), ABS EOSINOPHILS (X10^9/L), ABS LYMPHOCYTES (X10^9/L), ABS MONOCYTES (X10^9/L), and ABS NEUTROPHILS (X10^9/L) are presented.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: (X10^9/L)
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
(X10^9/L)
  ABS BASOPHILS (X10^9/L) | -0.00 (0.040) | 0.00 (0.035)
  ABS EOSINOPHILS (X10^9/L) | -0.01 (0.1) | 0.01 (0.115)
  ABS LYMPHOCYTES (X10^9/L) | -0.09 (0.535) | -0.03 (0.538)
  ABS MONOCYTES (X10^9/L) | 0.01 (0.134) | -0.00 (0.148)
  ABS NEUTROPHILS (X10^9/L) | 0.01 (1.542) | -0.10 (1.346)
  PLATELETS (X10^9/L) | -0.01 (44.126) | 1.82 (54.452)
  WBC (X10^9/L) | -0.09 (1.813) | -0.12 (1.614)

17. Secondary Outcome: Hematology - Hematocrit (Change From Baseline)
Description: A summary of a secondary safety outcome measure, Hematology - Hematocrit(HCT)(Change from Baseline), by treatment assigned, is shown for the safety population.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
percent | -0.58 (2.294) | -1.13 (3.093)

18. Secondary Outcome: Hematology - Hemoglobin (Change From Baseline)
Description: A summary of a secondary safety outcome measure, Hematology - Hemoglobin(HGB)(Change from Baseline), by treatment assigned, is shown for the safety population.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
g/dL | -0.18 (0.694) | -0.36 (0.854)

19. Secondary Outcome: Hematology - Red Blood Cell (Change From Baseline)
Description: A summary of a secondary safety outcome measure, Hematology - Red Blood Cell (RBC)(Change from Baseline), by treatment assigned, is shown for the safety population.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: x10^12/L
Arm/Group | Placebo | EMSAM
Number analyzed (Participants) | 156 | 152
x10^12/L | -0.04 (0.234) | -0.12 (0.313)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | EMSAM
Serious Adverse Events (participants affected / at risk) | 3/156 | 7/152
Other Adverse Events (participants affected / at risk) | 90/156 | 95/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=156) | EMSAM (N=152)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Loss of Consciousness (General disorders) | 1 (1) | 0 (0)
Mood Swings (Psychiatric disorders) | 1 (1) | 0 (0)
Orthstatic Hypotension (General disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Screaming (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 2 (2)
Syncope (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=156) | EMSAM (N=152)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (7) | 4 (4)
Agitation (Psychiatric disorders) | 3 (3) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Application Site Reaction (General disorders) | 34 (34) | 37 (37)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Dizziness (Nervous system disorders) | 7 (7) | 8 (8)
Fatigue (General disorders) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 26 (26) | 26 (26)
Insomnia (Psychiatric disorders) | 4 (4) | 9 (9)
Irritability (Psychiatric disorders) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (6)
Nausea (Gastrointestinal disorders) | 12 (12) | 11 (11)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 4 (4) | 7 (7)
Suicidal Ideation (Psychiatric disorders) | 4 (4) | 4 (4)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator is free to publish for their own research or publication objectives, provided that such does not disclose Confidential Information. At least 45 days prior the Investigator shall submit for Sponsor review. Sponsor will advise of revisions necessary to preserve confidential and proprietary information. The first publication of the results shall be a joint Multi-Center publication of results with the investigators from all study sites contributing data.